CLINICAL TRIAL: NCT07324161
Title: Efficacy and Safety of Repetitive Transcranial Magnetic Stimulation in the Treatment of Alzheimer's Disease and Exploration of Glymphatic Mechanisms
Brief Title: Efficacy and Safety of Transcranial Magnetic Stimulation in Treatment of Alzheimer's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: rTMS
Record Dates: First submitted 2025-12-24; First posted 2026-01-07 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer s Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS (Experimental)
  Interventions: Device: rTMS
- sham rTMS (Sham Comparator)
  Interventions: Device: sham rTMS

INTERVENTIONS:
Device: rTMS — Stimulation coil Cool-B65 A CO, positioning individualised, stimulation frequency 20Hz, stimulation intensity 100% of motor threshold, stimulation number 40 pulses/train, train interval 28s, 40 trains, 1600 total stimulation pulses, total stimulation time 20 min, treatment application once a day, continuous application for two weeks, 5 days a week.Consolidation therapy was also administered weekly for 6 months.
  Arms: rTMS
Device: sham rTMS — Stimulation coil Cool-B65 P CO, positioning individualised, stimulation frequency 20Hz, stimulation intensity 100% of motor threshold, stimulation number 40 pulses/train, train interval 28s, 40 trains, 1600 total stimulation pulses, total stimulation time 20 min, treatment application once a day, continuous application for two weeks, 5 days a week
  Arms: sham rTMS

SUMMARY:
This study is grounded in the regulatory mechanisms of the glymphatic system and applies repetitive transcranial magnetic stimulation (rTMS) to the treatment of Alzheimer's disease (AD). The clinical efficacy and safety of rTMS will be systematically evaluated. Furthermore, transcranial magnetic stimulation-evoked potentials (TMS-EEG) and functional near-infrared spectroscopy (fNIRS) will be employed to investigate, from the perspectives of synaptic plasticity and neurovascular coupling, the mechanisms by which rTMS influences glymphatic function. Collectively, this work aims to provide new insights into both the therapeutic effectiveness and the underlying mechanisms of rTMS in AD.

ELIGIBILITY:
Inclusion Criteria:

* Meets the 2018 NIA-AA diagnostic criteria for Alzheimer's disease (AD)
* Meets DSM-5 diagnostic criteria
* Mild to moderate disease severity (CDR Global Score 1 to 2)
* Evidence of AD pathology: positive amyloid PET OR positive cerebrospinal fluid (CSF) AD biomarkers OR positive plasma AD biomarkers

Exclusion Criteria:

* Contraindications to rTMS treatment
* Severe complications or immune diseases
* Unable to cooperate with study procedures
* History of epilepsy

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
MoCA Changes from baseline to post-treatment | Baseline vs 2 weeks and 6 months after treatment
  Montreal Cognitive Assessment (MoCA)

SECONDARY OUTCOMES:
CDR Changes from baseline to post-treatment | Baseline vs 2 weeks and 6 months after treatment
  Clinical Dementia Rating (CDR)
MMSE Changes from baseline to post-treatment | Baseline vs 2 weeks and 6 months after treatment
  Mini-Mental State Examination (MMSE)
NPI Changes from baseline to post-treatment | Baseline vs 2 weeks and 6 months after treatment
  Neuropsychiatric Inventory (NPI)
Neuropathological markers Change from baseline to post-treatment | Baseline vs 2 weeks and 6 months after treatment
  Aβ, tau, GFAP, NFL, VEGF
TMS-EEG Changes from baseline to post-treatment | Baseline vs 2 weeks and 6 months after treatment
  Concurrent transcranial magnetic stimulation and electroencephalography (TMS-EEG)

CONTACTS AND LOCATIONS:
Locations (1):
- rTMS, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No